CLINICAL TRIAL: NCT01143493
Title: The Role of Glucocorticoid Receptor SNPs in Receptor Function and Metabolic Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100130; 10-E-0130
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Glucose Homeostasis; Protein Metabolism; Lipid Metabolism; Respiratory Function; Connective Tissue Metabolism
Keywords: Genetic Polymorphism; Glucocorticoid; Health Volunteer; HV
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Carrier - Other
- Carrier hGR N363S Heterozygote
- Carrier hGR N363S Homozygote
- Carrier hGR9B A3669G Heterozygote
- Carrier hGR9B A3669G Homozygote
- Control

SUMMARY:
Background:

- Glucocorticoids are primary stress response hormones released from the adrenal gland when an individual is under stress. Chronic or ongoing elevation of these hormones due to prolonged stress or medical treatments can have numerous harmful effects. Researchers are interested in learning more about how these hormones affect cell growth, development, and death. To study glucocorticoid hormones, researchers plan to use the medication dexamethasone, which affects the parts of cells that respond to glucocorticoid hormones.

Objectives:

- To study glucocorticoid stress hormones in healthy individuals before and after receiving dexamethasone.

Eligibility:

* Healthy individuals at least 18 years of age.
* Participants must not be using certain medications that may affect the dexamethasone test, including hormonal contraception, steroid-based drugs, and some antidepressants.

Design:

* This study will require an initial screening visit and a second study visit. The visits are estimated to require about 1 to 2 hours of participation over a period of up to 14 days.
* Participants will be screened at visit 1 with a full physical examination and medical history, and an initial blood sample for testing.
* For visit 2, participants will be asked to abstain from all food and drinks except for water for 12 hours before the appointment, and will take one tablet of dexamethasone 9 hours before the appointment.
* Participants will have a second blood sample taken during visit 2, and will receive a snack after the blood is drawn.

DETAILED DESCRIPTION:
STUDY DESIGN:

This in vivo and in vitro observational gene association study will investigate the functional relevance of SNPs in the NR3C1 gene in selected populations. A subgroup of the EPR will be genotyped to identify novel SNPs in the NR3C1 gene. The most promising SNPs for functional relevance in in vitro assays will be examined. Individuals with and without functionally relevant, novel SNPs will be recruited for further study. In part 1, lymphocytes from these participants will be isolated, exposed ex vivo to corticosteroids, and gene expression profiles in response to this stimulus will be compared. In part 2, in vivo effect of these SNPs in steroid responsiveness will be evaluated by performing a modified low dose dexamethasone suppression test comparing by genotype. The study design is innovative as a gene association study in the sense that participants are recruited on the basis of genotype and then the phenotype of each participant is observed.

STUDY DURATION:

It is anticipated that the study will require 48 months to complete participants study visits.

PRIMARY OBJECTIVE:

Investigate in vivo the role of hGR SNPs (hGR9beta A3669B, hGR N363S) in steroid responsiveness by performing a modified dexamethasone suppression test and comparing responses by genotype.

SECONDARY OBJECTIVE:

Investigate the role of hGR SNPs (hGR9beta A3669B, hGR N363S) in human steroid responsiveness by comparing (across genotypes) gene expression profiles of isolated macrophages and lymphocytes exposed ex vivo to corticosteroids.

PRIMARY ENDPOINT:

Measure the change in serum cortisol levels after modified dexamethasone suppression test.

SECONDARY ENDPOINT:

Measure gene expression fold changes by microarray analysis after ex vivo glucocorticoid exposure of macrophages and lymphocytes; validation of affected RNA (elevated or decreased expression) through PCR analysis.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PART 1 AND 2:
* Male or female 18 years of age or older at the time of enrollment
* Must be a participant in the EPR study
* Are genotyped and determined to be heterozygote or homozygote carriers of one of the two hGR SNPs (hGR9B A3669G and hGR N363S) or are wild type at the SNP location
* Able to understand and provide written informed consent to participate in the study
* Able to travel to the CRU
* Willing and able to fast for periods of up to 12 hours during the study
* Healthy participants as defined by the International Red Cross guidelines (Healthy means that an individual feels well and can perform normal activities. If the individual has a chronic condition such as diabetes or high blood pressure, healthy also means that they are being treated and the condition is under control).

EXCLUSION CRITERIA:

Exclusion Criteria for Part 1

Participants with the following history will be excluded from part 1 of the study:

* Any glucocorticoid use within approximately 14 days of scheduled visit 1 including oral, inhaled, nasal sprays, and cream (dermal/mucosal)
* Pregnant or currently breastfeeding
* Planning to use certain medications because they can affect test results.
* Any condition that, in the investigator's opinion, places the participant at undue risk for complications.

Exclusion Criteria for Part 2

Participants with the following history will be excluded from part 2 of the study to avoid confounding the dexamethasone suppression test:

* Any glucocorticoid use within approximately 14 days of scheduled visit 2 including oral, inhaled, nasal sprays, and cream (dermal/mucosal)
* Pregnant or currently breastfeeding
* Currently enrolled in another clinical research study and/or is receiving an investigational agent for any reason
* Does not agree to take dexamethasone at scheduled time
* Planning to use certain medications such as corticosteroids, estrogens, or tetracyclines prior to the visit 2, because they can affect test results. If the participant is willing to withhold these medications for 14 days, then the participant will be allowed to participate in visit 2.

Participants with the following history will be excluded from part 2 of the study because the dexamethasone may cause potential harm to the participant:

* High blood pressure of 160/10 mm Hg or above.
* Active coronary artery disease (angina) or moderate to severe heart failure stage New York Heart Association III-IV
* Renal failure
* Glaucoma
* Uncontrolled psychiatric disorders such as bipolar disorder or schizoaffective disorder
* Active systemic fungal infection
* Prior hypersensitivity reaction to Dexamethasone
* Currently receiving treatment for cancer (certain cancers, like lung cancer make adrenocorticotropic hormone (ACTH), and all induce stress)
* Any condition that, in the investigator's opinion, places the participant at undue risk for complications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2010-09-30; Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Measure the change in serum cortisol levels after modified dexamethasone suppression test | baseline level in first visit, posttreatment level in second visit
  The null hypothesis for this endpoint (primary hypothesis for this study) is that there is no difference among genotypes in the change from baseline cortisol level. The two-sided alternative hypothesis is that there is a trend(homozygous wild-type to heterozygous to homozygous for the minor allele) in change from baseline.

SECONDARY OUTCOMES:
Measure gene expression fold changes by microarray analysis after ex vivo glucocorticoid exposure of macrophages and lymphocytes; validation of affected RNA (elevated or decreased expression) through PCR analysis. | The cells are cultured from blood drawn from participants at the first clinic visit.
  The secondary null hypotheses are that there are no differences among genotypes in fold-change for expression level (measured by RT-PCR for the genes selected by the microarray analysis as having differential expression), and the two-sided alternative is that there are trends.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Garantziotis, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. N Engl J Med. 2005 Oct 20;353(16):1711-23. doi: 10.1056/NEJMra050541. No abstract available. PMID 16236742
- [Background] DeRijk RH, Schaaf M, de Kloet ER. Glucocorticoid receptor variants: clinical implications. J Steroid Biochem Mol Biol. 2002 Jun;81(2):103-22. doi: 10.1016/s0960-0760(02)00062-6. PMID 12137800
- [Background] Huizenga NA, Koper JW, de Lange P, Pols HA, Stolk RP, Grobbee DE, de Jong FH, Lamberts SW. Interperson variability but intraperson stability of baseline plasma cortisol concentrations, and its relation to feedback sensitivity of the hypothalamo-pituitary-adrenal axis to a low dose of dexamethasone in elderly individuals. J Clin Endocrinol Metab. 1998 Jan;83(1):47-54. doi: 10.1210/jcem.83.1.4498. PMID 9435415